CLINICAL TRIAL: NCT02830074
Title: Does Treatment of Sleep-Disordered Breathing Improve Functional Outcomes in SCI
Brief Title: Treatment of Sleep-disordered Breathing in Patients With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2116-R; IRX002116A (Other Grant/Funding Number: VA)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Spinal Cord Injury; Sleep-disordered Breathing; Spinal Cord Disease; Multiple Sclerosis
Keywords: Sleep Apnea Syndromes; Spinal Cord Injuries; Sleep; Quality of life
MeSH Terms: conditions — Spinal Cord Injuries; Sleep Apnea Syndromes; Spinal Cord Diseases; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The BEST Program (Experimental): a combined sleep and PAP adherence program, called the BEST program (Best practices PAP + patient Education + ongoing Support and Training)
  Interventions: Behavioral: Best practices PAP + patient Education +ongoing Support and Training
- Sleep Education and standard SDB treatment (Active Comparator): This program includes non-directive sleep education plus standard treatment of SDB.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Best practices PAP + patient Education +ongoing Support and Training — This is a combined sleep and PAP adherence program, called the "BEST" program (Best practices PAP + Education + ongoing Support/Training
  Arms: The BEST Program
Behavioral: Sleep Education — This program includes non-directive sleep education plus standard treatment of SDB.
  Arms: Sleep Education and standard SDB treatment

SUMMARY:
Sleep-disordered breathing (SDB) remains under-treated in individuals living with spinal cord injuries and disorders (SCI/D). The investigators' aim is to test a program that addresses challenges and barriers to positive airway pressure (PAP) treatment of SDB among patients with SCI/D. The investigators anticipate that patients who receive this program will have higher rates of PAP use and will demonstrate improvements in sleep quality, general functioning, respiratory functioning and quality of life from baseline to 6 months follow up compared to individuals who receive a control program. This work addresses critical healthcare needs for patients with SCI/D and may lead to improved health and quality of life for these patients.

DETAILED DESCRIPTION:
This proposal aims to test the efficacy of a comprehensive approach to improving positive airway pressure (PAP) therapy acceptance and adherence and sleep quality among patients with SCI/D. The proposed study is very relevant to the mission of the VA in promoting optimal health for all Veterans, including those with disabilities. To this end, this study is a randomized controlled trial (RCT) comparing the efficacy of a combined sleep and PAP adherence program, called the "BEST" program (Best practices PAP + patient Education +ongoing Support and Training). The central aim of this proposal therefore is to test the efficacy between two PAP adherence programs. The study has two main aims. First, the investigators aim to test the efficacy of the educational program in improving adherence to PAP therapy for the first 6 months of use (with data available for some subjects for up to 12 months). Second, the investigators will evaluate the impact of the program on sleep quality and on three key areas of function: general functioning (using measures specific to SCI/D patients), respiratory functioning (via spirometry) and quality of life (assessed with measures appropriate for use with patients having limited mobility) over the 3-month intervention period. The investigators will also explore whether the intervention is more effective for some subgroups of patients than others. The proposed work is very relevant to VA's patient care mission, addressing a critical need for patients who suffer from disparity in access to high quality care because of their disabilities. The investigators anticipate that the investigators' work will yield significant new knowledge that improves the health and quality of life for Veterans living with SCI/D.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic SCI/D (>3 months post injury)
* American Spinal Injury Association (ASIA) classification A-D (i.e., excluding those with no evidence of a neurologic deficit based on ASIA classification).

Exclusion Criteria:

* Patients receiving mechanical ventilation
* already using PAP for SDB at optimal compliance
* A clinical contraindication that prevents PAP use.
* recent health event that may affect sleep, e.g.:

  * CVA
  * acute MI
  * recent surgery or hospitalization
* alcohol or substance abuse (<90 days sobriety)
* self-described as too ill to engage in study procedures
* unable to provide self-consent for participation (e.g., due to dementia)
* the investigators will offer to re-contact patients 90 days after a health event or after 90 days of sobriety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M S Badr, MD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badr AN, Zeineddine S, Salloum A, Pandya N, Mitchell MN, Sankari A, Munoz ID, Badr MS, Martin JL, Kelly MR. Sleep and daytime function in people with spinal cord injury. J Clin Sleep Med. 2025 Nov 1;21(11):1903-1909. doi: 10.5664/jcsm.11804. PMID 40590079
- [Derived] Badr MS, Martin JL, Sankari A, Zeineddine S, Salloum A, Henzel MK, Strohl K, Shamim-Uzzaman A, May AM, Fung CH, Pandya N, Carroll S, Mitchell MN. Intensive support does not improve positive-airway pressure use in spinal cord injury/disease: a randomized clinical trial. Sleep. 2024 May 10;47(5):zsae044. doi: 10.1093/sleep/zsae044. PMID 38422375
- [Derived] Kelly MR, Zeineddine S, Mitchell MN, Sankari A, Pandya N, Carroll S, Shamim-Uzzaman QA, Salloum A, Badr MS, Martin JL. Insomnia severity predicts depression, anxiety, and posttraumatic stress disorder in veterans with spinal cord injury or disease: a cross-sectional observational study. J Clin Sleep Med. 2023 Apr 1;19(4):695-701. doi: 10.5664/jcsm.10410. PMID 36661092

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 Participants started the study and out of those 73 participants only 63 were randomized. Therefore, only 63 participants out of 73 were eligible to be randomized ( 1 ineligible, 3 withdraw, 3 passive withdraw, 2 AHI<5, 1 Pilot).
Period: Overall Study
Arm/Group | The BEST Program | Sleep Education and Standard SDB Treatment
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- The BEST Program: a combined sleep and PAP adherence program, called the ?BEST? program (Best practices PAP + patient Education + ongoing Support and Training)
  Best practices PAP + patient Education +ongoing Support and Training: This is a combined sleep and PAP adherence program, called the "BEST" program (Best practices PAP + Education + ongoing Support/Training
- Total: Total of all reporting groups
Arm/Group | The BEST Program | Sleep Education and Standard SDB Treatment | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.63 (10.02) | 59.80 (10.44) | 60.73 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 29 | 29 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 16 | 15 | 31
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 31 | 63
Apnea Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events/hr] — Apnea Hypopnea Index (AHI) is an index measure of the number of apneas and hypopneas per hour. While there is no maximum value, 0-5 is considered normal, 5-15 is considered mild sleep disordered breathing, and anything greater or equal to 15 is considered severe sleep disordered breathing.
  events/hr | 30.19 (22.92) | 30.32 (24.87) | 30.25 (23.71)

OUTCOME MEASURES:

1. Primary Outcome: PAP Adherence
Description: Number of nights positive airway pressure (PAP) was used >=4 hours during the first 90 days measured by remote monitoring. Scores range from 0 to 90 days. Higher scores indicate better outcome.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: nights
Groups:
- Sleep Education and Standard Sleep-disordered Breathing Treatment: This program includes non-directive sleep education plus standard treatment of sleep-disordered breathing .
  Sleep Education: This program includes non-directive sleep education plus standard treatment of sleep-disordered breathing .
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing Treatment
Number analyzed (Participants) | 32 | 31
nights | 22.03 (24.74) | 18.54 (24.67)

2. Primary Outcome: Subjective Sleep Quality Was Measured by The Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is an 18-item questionnaire that assesses sleep quality and disturbances over the past month. The PSQI is sensitive for distinguishing normal and abnormal sleepers and has good test-retest reliability. The investigators will use the 3-factor scoring, which has been shown to have superior psychometric properties. This will be used as the main independent measure of sleep quality.
  The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality
Time Frame: 90 days
Population: 63 were randomized, 60 participants were analyzed for the 90 day period, due to missing data on study forms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing Treatment
Number analyzed (Participants) | 30 | 30
units on a scale | 6.96 (4.12) | 9.1 (4.97)

3. Secondary Outcome: Quality of Life Was Measured by WHO-QOL BREF Questionnaire
Description: The questionnaire is composed of four domains: physical health, psychological health, social relationships and environment. It also includes one question on overall quality of life and one on general health. Importantly, items on this scale are not dependent on mobility, which is unlikely to change in patients with Spinal Cord Injury/Disease as a result of improved sleep. The WHOQOL-BREF scores correlate highly (.89 or above) with WHOQOL-100 scores, and demonstrate good discriminant validity, content validity, internal consistency and test-retest reliability. The four WHOQOL-BREF domain scores will be used as main outcome measure. The WHOQOL-BREF measures quality of life across 4 domains. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval, higher score correspond to greater perceived quality of life
Time Frame: 90 days
Population: 63 were randomized, 62 participants were analyzed for the 90 day period, due to missing data on study forms.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sleep Education and Standard Sleep-disordered Breathing (SDB) Treatment: This program includes non-directive sleep education plus standard treatment of SDB.
  Sleep Education: This program includes non-directive sleep education plus standard treatment of SDB.
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing (SDB) Treatment
Number analyzed (Participants) | 31 | 31
units on a scale
  WHO-QOL phys | 60.13 (21.37) | 54.72 (22.08)
  WHO-QOL psych | 69.22 (14.69) | 62.90 (19.64)
  WHO-QOL Soc | 63.70 (24.39) | 57.52 (23.20)
  WHO-QOL ENV | 74.09 (12.66) | 69.75 (18.40)

4. Secondary Outcome: Respiratory Function: Spirometry and Respiratory Muscle Force
Description: Spirometry is a simple bedside test used to evaluate lung function. Key spirometry values include forced vital capacity (FVC) and forced expiratory volume over 1 second (FEV1) and the absolute FEV1/FVC ratio. If the FVC and FEV1 are decreased, the absolute FEV1/FVC ratio distinguishes between obstructive and restrictive impairments. A normal absolute FEV1/FVC ratio suggest that restrictive ventilatory impairment may be present, and a reduced FEV1 and absolute FEV1/FVC ratio indicates an obstructive ventilator pattern. The investigators will use supine FVC and maximal inspiratory pressure (MIP) as the key outcome measures for respiratory function for this study, as these are the most representative of respiratory functioning during sleep.
  The normal value for the FEV1/FVC ratio is above 0.75. Values lower than 0.70 are suggestive of airflow limitation with an obstructive pattern whilst in restrictive lung diseases, this ratio is normal or high.
Time Frame: 90 days
Population: 63 were randomized, 60 participants were analyzed for the 90 day period, due to missing data on study forms.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing (SDB) Treatment
Number analyzed (Participants) | 30 | 30
ratio | 3.38 (1.04) | 3.20 (0.97)

5. Secondary Outcome: Functional Status Was Measured by CHART Questionnaire.
Description: The CHART is a measure of overall function. The scale is divided into five separate domain scores: Physical, Cognitive, Mobility, Occupation, and Social integration.
  Each of the five domains scored from 0-100. higher number indicates better outcome.
Time Frame: 90 days
Population: 63 were randomized, 62 participants were analyzed for the 90 day period, due to missing data on study forms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing (SDB) Treatment
Number analyzed (Participants) | 31 | 31
units on a scale
  Physical | 79.09 (31.02) | 82.70 (31.39)
  Cognitive | 70.70 (23.90) | 78.83 (22.44)
  Mobility | 82.20 (19.64) | 78.17 (24.33)
  Occupation | 48.98 (31.39) | 38.90 (33.76)
  Social integration | 79 (23.64) | 66.80 (29.42)

6. Secondary Outcome: Depressive Symptom Severity
Description: The Patient Health Questionnaire-9 (PHQ-9) is a 9-item depression module in the PHQ (a self-administered diagnostic instrument for common mental disorders) which is part of the Primary Care Evaluation of Mental Disorders (PRIME-MD) suite of evaluation tools. The PHQ-9 aligns to the DSM-IV diagnostic criteria for depression and is widely used to screen for depression across VA. The PHQ-9 total score will be used to measure depressive symptom severity as an outcome.
  As a severity measure, the PHQ-9 score can range from 0 to 27. Higher the value, worse the outcome.
Time Frame: 90 days
Population: 63 were randomized, 62 participants were analyzed for the 90 day period, due to missing data on study forms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing (SDB) Treatment
Number analyzed (Participants) | 31 | 31
units on a scale | 5.03 (5.89) | 8.38 (6.44)

7. Secondary Outcome: Fatigue Symptoms
Description: The Flinders Fatigue Scale (FFS) is a 7-item fatigue rating scale used to measure general symptoms of fatigue. The FFS total score will be used as an outcome measure.
  Total fatigue scores range from 0 to 31, with higher scores indicating greater fatigue.
Time Frame: 90 days
Population: 63 were randomized, 62 participants were analyzed for the 90 day period, due to missing data on study forms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing (SDB) Treatment
Number analyzed (Participants) | 31 | 31
units on a scale | 9.61 (8.46) | 12.12 (9.33)

8. Secondary Outcome: Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire that quantifies daytime sleepiness, with higher scores indicating increased daytime hypersomnolence The ESS is ranging from 0 to 24. higher scores indicate more sleepiness
Time Frame: 90 days
Population: 63 were randomized, 62 participants were analyzed for the 90 day period, due to missing data on study forms
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | The BEST Program | Sleep Education and Standard Sleep-disordered Breathing (SDB) Treatment
Number analyzed (Participants) | 31 | 31
units on a scale | 4.58 (4.94) | 6.48 (4.13)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | The BEST Program | Sleep Education and Standard SDB Treatment
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT02830074/Prot_002.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT02830074/SAP_000.pdf
  • Informed Consent Form (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT02830074/ICF_001.pdf